CLINICAL TRIAL: NCT02708095
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel- Group, Phase 2 Study of Baricitinib in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: A Study of Baricitinib (LY3009104) in Participants With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16270; I4V-MC-JAHH (Other: Eli Lilly and Company); 2015-004404-35 (EudraCT Number)
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2017-12

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 mg Baricitinib (Experimental): Participants received 2 (milligrams) mg of Baricitinib tablet orally once a day for 24 weeks.
  Interventions: Drug: Baricitinib
- 4 mg Baricitinib (Experimental): Participants received 4 mg of Baricitinib tablet orally once a day for 24 weeks.
  Interventions: Drug: Baricitinib
- Placebo (Placebo Comparator): Participants received Placebo orally once daily (QD) for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: 2 mg Baricitinib; 4 mg Baricitinib
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of the study drug known as baricitinib in participants with systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* Have received a diagnosis of SLE at least 24 weeks prior to screening, meeting the American College of Rheumatology (ACR) 1982 revised criteria OR the 2012 Systemic Lupus Erythematosus International Collaborating Clinics (SLICC) criteria.
* Have a positive antinuclear antibody (ANA) (titer ≥1:80) and/or a positive anti-double-stranded deoxyribonucleic acid (dsDNA) as assessed by a central laboratory at screening.
* Have a SLEDAI-2K score ≥4 based on clinical symptoms (not including lab values) at randomization.
* Have active arthritis and/or active rash as defined by the SLEDAI-2K at randomization.

Exclusion Criteria:

* Have active severe lupus nephritis.
* Have active severe central nervous system (CNS) lupus.
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data.
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection.
* Are currently receiving oral corticosteroids at doses >20-milligrams per day of prednisone (or equivalent) or have adjusted the dose of corticosteroids within 2 weeks of planned randomization.
* Have started treatment with or adjusted the dose of nonsteroidal anti-inflammatory drugs (NSAIDs) (for which the NSAID use is intended for treatment of signs and symptoms of SLE) within 4 weeks of planned randomization.
* Have started treatment with or adjusted the dose of an antimalarial within 12 weeks of planned randomization.
* Have started treatment with or adjusted the dose of an immunosuppressant within 12 weeks of planned randomization.
* Have received cyclophosphamide (or any other cytotoxic agent) within 12 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (77):
- United States (27):
  - University of Arizona, Tucson, Arizona
  - Wallace Rheumatic Study Center, Beverly Hills, California
  - Medvin Clinical Research, Covina, California
  - TriWest Research Assocaites, El Cajon, California
  - University of California, La Jolla, California
  - Desert Medical Advances, Palm Desert, California
  - Inlande Rheumatology Clinical Trials, Upland, California
  - Denver Arthritis Center, Denver, Colorado
  - New Horizon Research Center, Miami, Florida
  - West Broward Rheumatology Associates, Inc, Tamarac, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Kansas City Internal Medicine Research, Overland Park, Kansas
  - The Arthritis & Diabetes Clinic Inc., Monroe, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Clayton Medical Research, St Louis, Missouri
  - Arthritis Consultants, St Louis, Missouri
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - North Shore University Hospital at Great Neck, Great Neck, New York
  - The Ohio State University, Columbus, Ohio
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Arthritis & Rheumatology Center of Oklahoma PLLC, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - The Oklahoma Center For Arthritis Therapy, Tulsa, Oklahoma
  - East Penn Rheumatology, Bethlehem, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - Accent Clinical Research Professionals, LLC, Allen, Texas
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Autonoma de Buenos Aire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pessac
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
- Japan (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asahikawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chūōku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamamatsu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Itabashi-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kawagoe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kita-gun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitakyushu
  - Meguro-kuFor additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meguro-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōmura
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sasebo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sendai
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zapopan
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bytom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nadarzyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Świdnik
- Puerto Rico (3):
  - Office: Perez-De Jesus, Amarilis, Caguas
  - Mindful Medical Research, San Juan
  - Latin Clinical Trial Center, Santurce
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galati
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gwangju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badalona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vigo
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei

REFERENCES:
- [Derived] Dorner T, Tanaka Y, Dow ER, Koch AE, Silk M, Ross Terres JA, Sims JT, Sun Z, de la Torre I, Petri M. Mechanism of action of baricitinib and identification of biomarkers and key immune pathways in patients with active systemic lupus erythematosus. Ann Rheum Dis. 2022 Aug 11;81(9):1267-1272. doi: 10.1136/annrheumdis-2022-222335. PMID 35609978
- [Derived] Dorner T, van Vollenhoven RF, Doria A, Jia B, Ross Terres JA, Silk ME, de Bono S, Fischer P, Wallace DJ. Baricitinib decreases anti-dsDNA in patients with systemic lupus erythematosus: results from a phase II double-blind, randomized, placebo-controlled trial. Arthritis Res Ther. 2022 May 16;24(1):112. doi: 10.1186/s13075-022-02794-x. PMID 35578304
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Wallace DJ, Furie RA, Tanaka Y, Kalunian KC, Mosca M, Petri MA, Dorner T, Cardiel MH, Bruce IN, Gomez E, Carmack T, DeLozier AM, Janes JM, Linnik MD, de Bono S, Silk ME, Hoffman RW. Baricitinib for systemic lupus erythematosus: a double-blind, randomised, placebo-controlled, phase 2 trial. Lancet. 2018 Jul 21;392(10143):222-231. doi: 10.1016/S0140-6736(18)31363-1. PMID 30043749
- See also: Click here for more information about this study: A Study of Baricitinib (LY3009104) in Participants With Systemic Lupus Erythematosus (SLE) — http://www.lillytrialguide.com/en-US/studies/lupus/JAHH#?postal=

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Started | 105 | 105 | 104
Received at Least 1 Dose of Study Drug | 105 | 105 | 104
Completed | 83 | 86 | 86
Not Completed | 22 | 19 | 18
Not completed — Adverse Event | 4 | 10 | 11
Not completed — Lack of Efficacy | 9 | 3 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Physician Decision | 2 | 3 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- 2 mg Baricitinib: Participants received 2 mg of Baricitinib tablet orally once a day for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib | Total
Number analyzed (Participants) | 105 | 105 | 104 | 314
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.9 (12.8) | 43.2 (11.0) | 45.0 (12.4) | 44.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 96 | 99 | 294
  Male | 6 | 9 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 32 | 32 | 102
  Not Hispanic or Latino | 52 | 62 | 60 | 174
  Unknown or Not Reported | 15 | 11 | 12 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 6 | 10 | 25
  Asian | 20 | 20 | 20 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 9 | 7 | 21
  White | 71 | 68 | 65 | 204
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 6 | 5 | 6 | 17
  Argentina | 9 | 12 | 7 | 28
  Austria | 3 | 2 | 3 | 8
  South Korea | 1 | 2 | 3 | 6
  Romania | 4 | 2 | 7 | 13
  United States | 31 | 34 | 30 | 95
  Japan | 13 | 10 | 10 | 33
  Taiwan | 6 | 7 | 5 | 18
  Poland | 13 | 10 | 9 | 32
  Mexico | 11 | 8 | 14 | 33
  France | 2 | 7 | 7 | 16
  Spain | 6 | 6 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Remission of Arthritis and/or Rash Defined by the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K)
Description: Participants were defined as responder as follows using SLEDAI-2K definitions of arthritis and rash. If only arthritis is present at baseline, then arthritis must be absent at Week 24 to meet the primary endpoint. If only rash is present at baseline, then rash must be absent at Week 24 to meet the primary endpoint. If both arthritis and rash are present at baseline, then the primary endpoint is met if either arthritis, or rash, or both arthritis and rash are absent at Week 24.
Time Frame: Week 24
Population: All randomized participants who received at least 1 dose of study drug with baseline and post-baseline values at the specified time point for remission of arthritis and/or rash.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 105 | 105 | 104
Percentage of Participants | 53.3 | 58.1 | 67.3
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.392, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.73 to 2.27]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.041, Regression, Logistic; Odds Ratio (OR) = 1.84, 95% CI 2-sided [1.02 to 3.29]

2. Secondary Outcome: Percentage of Participants Who Achieve SLE Responder Index 4 (SRI-4) Response
Description: SRI-4 response is defined as: 1) Reduction of ≥4 points from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score; 2) no new British Isles Lupus Assessment Group (BILAG) A or no more than 1 new BILAG B disease activity scores; and 3) no worsening (defined as an increase of ≥0.3 points [10 mm] from baseline) in Physician's Global Assessment of Disease Activity. The SRI-4 is a composite index used to assess disease activity in SLE. SLEDAI-2K assessment consists of 24 items with total score of 0 to 105, with higher scores representing increased disease activity. BILAG Index: assessing clinical signs, symptoms, or laboratory parameters related to SLE, divided into 9 organ systems. For each organ system: A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected. PGA is a visual analog scale scored from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe).
Time Frame: Week 24
Population: All randomized participants who received at least 1 dose of study drug with baseline and post-baseline values at the specified time point for SRI-4 response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 105 | 105 | 104
Percentage of Participants | 47.6 | 51.4 | 64.4
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.440, Regression, Logistic; Odds Ratio, log = 1.25, 95% CI 2-sided [0.71 to 2.19]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.015, Regression, Logistic; Odds Ratio (OR) = 2.04, 95% CI 2-sided [1.15 to 3.62]

3. Secondary Outcome: Change From Baseline in SLEDAI-2K Score
Description: SLE Disease Activity Index 2000 (SLEDAI-2K) score is a weighted, cumulative index of lupus disease activity. SLEDAI-2K is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with baseline of response, region, baseline disease activity (SLEDAI-2K <10, >=10), baseline anti-dsDNA status (positive, negative), treatment, time, treatment*time (type III sum of squares).
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug with baseline and post-baseline values at the specified time point for SLEDAI-2K.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 86 | 88 | 86
Units on a scale | -3.82 (0.352) | -4.07 (0.356) | -4.39 (0.353)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.600, Mixed Models Analysis; LS Mean Difference (Final Vaules) = -0.26, 95% CI 2-sided [-1.23 to 0.71]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.243, Mixed Models Analysis; LS Mean Difference (Final Vaules) = -0.58, 95% CI 2-sided [-1.55 to 0.39]

4. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity
Description: The Patient's Global Assessment of Disease Activity is a single-item, patient reported scale developed for the assessment of the patient's overall rating of their disease activity due to SLE. The scale measures disease activity through a 5 point Likert scale ranging from 0 ("No disease activity") to 4 ("Severe disease activity") at its worst over the past 7 days. LS mean was determined by MMRM model with baseline of response, region, baseline disease activity (SLEDAI-2K <10, >=10), baseline anti-dsDNA status (positive, negative), treatment, time, treatment*time (type III sum of squares).
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least 1 dose of study drug with baseline and post-baseline values at the specified time point for Patient's Global Assessment of Disease Activity.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 84 | 86 | 86
Units on a scale | -0.67 (0.105) | -0.83 (0.107) | -1.00 (0.105)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.285, Mixed Models Analysis; LS Mean Difference (Final Vaules) = -0.16, 95% CI 2-sided [-0.45 to 0.13]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.026, Mixed Models Analysis; LS Mean Difference (Final Vaules) = -0.33, 95% CI 2-sided [-0.62 to -0.04]

5. Secondary Outcome: Population Pharmacokinetics (PK): Area Under the Concentration-Time Curve of Baricitinib at Steady State (AUCτ, ss)
Description: Plasma samples for pharmacokinetic (PK) analysis were obtained in week 0, week 4, week 8, week 16 and 24. AUC takes all time points post dose into account and one value is reported.
Time Frame: Week (Wk) 0: 15-30 minutes (min) postdose; Wk 4: Predose, 1.5 - 4 hour (hr) postdose; Wk 8: 1 - 3 hr postdose; Wk 16: Predose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK (pharmacokinetics) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 104 | 104
nanogram*hour per milliliter (ng*h/mL) | 265 (55) | 569 (50)

6. Secondary Outcome: Population Pharmacokinetics (PK): Maximum Observed Drug Concentration at Steady State (Cmax,ss)
Description: Plasma samples for pharmacokinetic (PK) analysis were obtained in week 0, week 4, week 8, week 16 and 24. Cmax takes all time points post dose into account and one value is reported.
Time Frame: as for outcome 5
Population: All randomized participants who received at least one dose of study drug and had evaluable PK (pharmacokinetics) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 104 | 104
nanogram per milliliter (ng/mL) | 29.0 (30) | 59.2 (24)

ADVERSE EVENTS:
Time Frame: Up to 32 weeks
Description: All randomized participants who received at least 1 dose of study drug. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/105 | 0/104
Serious Adverse Events (participants affected / at risk) | 5/105 | 11/105 | 10/104
Other Adverse Events (participants affected / at risk) | 27/105 | 36/105 | 32/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=105) | 2 mg Baricitinib (N=105) | 4 mg Baricitinib (N=104)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0/99 (0) | 1/96 (1) | 0/99 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0/99 (0) | 1/96 (1) | 0/99 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=105) | 2 mg Baricitinib (N=105) | 4 mg Baricitinib (N=104)
Pharyngitis (Infections and infestations) | 3 (3) | 6 (6) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 7 (7) | 8 (8)
Urinary tract infection (Infections and infestations) | 11 (15) | 10 (12) | 9 (15)
Viral upper respiratory tract infection (Infections and infestations) | 4 (5) | 10 (13) | 10 (12)
Headache (Nervous system disorders) | 3 (3) | 6 (8) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-12-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT02708095/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT02708095/SAP_001.pdf